CLINICAL TRIAL: NCT07119710
Title: Improving Quality of Life in Persons Living in Rural Texas
Brief Title: Telehealth to Improve Quality of Life in Persons Living in Rural Texas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TexasTechU3
Record Dates: First submitted 2025-05-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Issue; Quality of Life
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavior Therapy (Experimental): Cognitive Behavior Therapy is an evidence-based practice for mental health conditions and has been shown in numerous studies around the world to be effective.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Cognitive Behavior Therapy plus 2 check-in calls a week (Experimental): This arm will provide the same as the first with the addition of twice-weekly check-in calls between sessions.
  Interventions: Behavioral: Cognitive Behavioral therapy with 2 check in calls

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Individual tele-therapy 12-16 weeks
  Arms: Cognitive Behavior Therapy
Behavioral: Cognitive Behavioral therapy with 2 check in calls — Cognitive Behavioral therapy with 2 calls a week
  Arms: Cognitive Behavior Therapy plus 2 check-in calls a week

SUMMARY:
The overarching goal of this project is to evaluate a current evidence-based practice, Cognitive Behavioral Therapy, for mental health conditions against Cognitive Behavioral Therapy plus two check-in calls a week for adults living in rural Texas.

DETAILED DESCRIPTION:
This two-armed study, for adults living in rural Texas, aims to evaluate current evidence-based practice, Cognitive Behavioral Therapy, for mental health conditions against Cognitive Behavioral Therapy plus two check-in calls a weel.

ELIGIBILITY:
Inclusion Criteria:

* family caregiver of person with all forms of dementia

Exclusion Criteria:

* not in another clinical intervention

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Pre-death grief (PG-12) | Baseline Weekly before the intervention 1 Month following the intervention 3 Months following the intervention 6 months following the intervention
  PG-12 is a questionnaire used to assess grief experiences before the death of a person will a life limiting illness. It is designed for caregivers of individuals with life limiting illnesses, including those with cancer or dementia. The PG-12 helps identify individuals at risk for prolonged grief disorder (PGD) and can be used in conjunction with other assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Garrison Institute on Aging, Lubbock, Texas, United States